CLINICAL TRIAL: NCT05359276
Title: Acid Sphingomyelinase Deficiency (ASMD): Data Analysis of Adult and Pediatric Patients on Early Access to Olipudase Alfa in France
Brief Title: Data Analysis of Adult and Pediatric Participants With Acid Sphingomyelinase Deficiency (ASMD) on Early Access to Olipudase Alfa in France
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17422
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Acid Sphingomyelinase Deficiency (ASMD)
MeSH Terms: conditions — Niemann-Pick Diseases | interventions — olipudase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with a confirmed diagnosis of ASMD under early access to olipudase alfa in France
  Interventions: Drug: Olipudase alfa

INTERVENTIONS:
Drug: Olipudase alfa — GZ402665

SUMMARY:
Primary Objective:

To describe the lung, spleen and liver outcomes of olipudase alfa

Secondary Objectives:

* To describe the patient's characteristics
* To describe conditions of olipudase alfa use
* To describe safety data related to the use of olipudase alfa
* To describe complementary effectiveness outcomes parameters

DETAILED DESCRIPTION:
Approximate duration of enrollment: 30 months

Total study duration: approximately 30 months

This is a national, multicenter observational retrospective and prospective cohort data collection study. Retrospective is defined as collection of data from all patients, including deceased patients, who were already on early access olipudase alfa in France before the start of this study.

ELIGIBILITY:
Inclusion Criteria:

* The patient, or the patient's parent(s)/guardian(s), has signed written informed consent.
* Patients with a confirmed diagnosis of ASMD under early access to olipudase alfa in France (ie, nominative compassionate use, pre marketing authorization early access, post marketing authorization early access).
* The patient has documented deficiency of acid sphingomyelinase in peripheral leukocytes, lymphocytes, or cultured fibroblasts.
* Male and female patients of all ages.

Exclusion Criteria:

* The patient or legal guardian(s) who has not received information notice or who opposes to data collection.
* Patient who died before study initiation and who was opposed to data collection for research purpose when he/she was alive.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of ASMD under early access to olipudase alfa in France (with a written informed consent)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary function diffusion capacity of lung for carbon monoxide (DLco) | From baseline to 24 months
Change in spleen size | From baseline to 24 months
Change in liver size | From baseline to 24 months

SECONDARY OUTCOMES:
Baseline patient characteristics | At baseline
  Demographic and baseline data [age, gender, weight, phenotype and genotype of ASMD, acid sphingomyelinase activity in peripheral leukocytes, lymphocytes, or cultured fibroblasts, age at diagnosis, age at first symptom onset, history of splenectomy (month/year), habits (i.e., smoking, alcoholism), known metabolic conditions or diseases (obesity, diabetes, familial dyslipidemias), known respiratory diseases; known hepatic diseases; others)]
Condition of olipudase alfa use | From baseline up to 3 years
  Conditions of olipudase alfa use (time to reach maximum dose [3 mg/kg] or the maximum tolerated dose for the patient, center profile, treater specialty, need of a premedication before the infusion [if yes, precise], treatment duration [start and end dates], treatment discontinuation [Yes/No] and reason of treatment discontinuation if any)
Safety: AE | From baseline up to 3 years
  Number of Participants with Adverse events (AE) including infusion-associated reactions
Safety: immunogenicity | From baseline up to 3 years
  Immune response assessments (antibodies anti-olipudase alfa IgG)
Complementary effectiveness: change in pulmonary function DLco | From baseline to 12 months and 36 months
Complementary effectiveness: change in spleen size | From baseline to 12 months and 36 months
Complementary effectiveness: change in liver size | FFrom baseline to 12 months and 36 months
Change in interstitial pulmonary infiltration based on lung imaging (thoracic CT-scan) | From baseline to 12 months and 24 months
Change in platelet count | From baseline at 3, 6, 9, 12, 24 months and every year up to 3 years
Change in biomarkers (chitotriosidase and lysosphingomyelin) plasma levels | From baseline at 3, 6, 9, 12 months and every year up to 3 years
Change in liver function | From baseline at 3, 6, 9, 12, 24 months and every year up to 3 years
  Alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total and direct bilirubin
Change in lipid profile | From baseline at 3, 6, 9, 12, 24 months and every year up to 3 years
  total cholesterol, high density lipoprotein (HDL) and low density lipoprotein (LDL) cholesterol
Change in growth curve for pediatric patient | From baseline at 6, 12, 24 months and every year up to 3 years
Change in weight | From baseline to 12 months and 36 months
Number of Participants with Evolution of Comorbidities | From baseline to 12 months, 24 months and 36 months
  Number of participants with evolution of comorbidities will be assessed by grade, attenuation or disappearance/absence

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site in France, France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org